CLINICAL TRIAL: NCT03234907
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Examine the Efficacy and Safety of Intravenous Vedolizumab (300 mg) Infusion Treatment in Chinese Subjects With Moderately to Severely Active Crohn's Disease
Brief Title: Vedolizumab Intravenous (IV) Compared to Placebo in Chinese Participants With Crohn's Disease.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Vedolizumab-3034; U1111-1195-3932 (Other: World Health Organization)
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Results first posted 2022-09-21 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Crohn's Disease
Keywords: Drug therapy
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Induction Phase: Placebo (Placebo Comparator): Placebo, IV, infusion, once at Weeks 0, 2, and 6 in the Induction Phase.
  Interventions: Drug: Vedolizumab IV
- Induction Phase: Vedolizumab 300 mg (Experimental): Vedolizumab 300 milligram (mg), IV infusion, once at Weeks 0, 2, and 6 in the Induction Phase.
  Interventions: Drug: Placebo
- Maintenance Phase: Induction Placebo to Placebo Q4W (Placebo Comparator): Participants who received placebo in the Induction Phase and achieved clinical response at Week 10 continued to receive placebo in the Maintenance Phase. Vedolizumab placebo-matching, IV infusion, once every 4 weeks (Q4W), from Week 14 to Week 58.
  Interventions: Drug: Vedolizumab IV; Drug: Placebo
- Maintenance Phase: Induction Placebo to Vedolizumab 300 mg Q4W (Experimental): Participants who received placebo in the Induction Phase and did not achieve clinical response at Week 10 received vedolizumab in the Maintenance Phase. Vedolizumab 300 mg, IV infusion, Q4W, from Week 14 to Week 58.
  Interventions: Drug: Vedolizumab IV
- Maintenance Phase: Induction Vedolizumab 300 mg to Vedolizumab 300 mg Q8W (Experimental): Participants who received vedolizumab in the Induction Phase and achieved clinical response at Week 10 continued to receive vedolizumab in the Maintenance Phase. Vedolizumab 300 mg, IV infusion, once every 8 weeks (Q8W), at Weeks 14, 22, 30, 38, 46 and 54 and vedolizumab placebo-matching, IV infusion, Q8W, at Weeks 18, 26, 34, 42, 50 and 58 to maintain double-blind.
  Interventions: Drug: Placebo
- Maintenance Phase: Induction Vedolizumab 300 mg to Vedolizumab 300 mg Q4W (Experimental): Participants who received vedolizumab in the Induction Phase and did not achieve clinical response at Week 10 received vedolizumab in the Maintenance Phase. Vedolizumab 300 mg, IV infusion, Q4W, from Week 14 to Week 58.
  Interventions: Drug: Vedolizumab IV

INTERVENTIONS:
Drug: Vedolizumab IV — Vedolizumab IV infusion
  Arms: Induction Phase: Placebo; Maintenance Phase: Induction Placebo to Placebo Q4W; Maintenance Phase: Induction Placebo to Vedolizumab 300 mg Q4W; Maintenance Phase: Induction Vedolizumab 300 mg to Vedolizumab 300 mg Q4W
Drug: Placebo — Vedolizumab placebo-matching
  Arms: Induction Phase: Vedolizumab 300 mg; Maintenance Phase: Induction Placebo to Placebo Q4W; Maintenance Phase: Induction Vedolizumab 300 mg to Vedolizumab 300 mg Q8W

SUMMARY:
The purpose of this study is to assess the safety and efficacy of vedolizumab intravenous (IV) infusion as induction treatment in Chinese participants with moderately to severely active Crohn's disease (CD) at Week 10.

DETAILED DESCRIPTION:
The drug being tested in this study is called vedolizumab. Vedolizumab will be administered as an intravenous (IV) infusion in Chinese participants. This study will investigate the efficacy and safety of vedolizumab IV as induction and maintenance therapy in participants with moderately to severely active Crohn's Disease (CD).

The study will enroll approximately 300 moderately to severely active Chinese patients with CD.

Induction Phase: participants will be randomized 2:1 to receive:

* Vedolizumab IV 300 mg
* Placebo IV

Participants will receive vedolizumab 300 mg or matching placebo, intravenous (IV) infusion at Weeks 0, 2, and 6 in the induction phase. At Week 10, participants will be assessed for clinical response. Results of Week 10 clinical response will determine the treatment pathway in the maintenance phase.

Maintenance Phase: participants who achieved clinical response at Week 10 will continue to receive the same treatment as they received in Induction Phase; every 8 weeks (Q8W) starting at Week 14. Participants who received vedolizumab IV or placebo in the Induction Phase and did not achieve clinical response at Week 10 will receive vedolizumab every 4 weeks (Q4W) starting at Week 14.

This multi-center trial will be conducted in China. The overall time to participate in this study is 60 weeks. Participants will make multiple visits to the clinic, and will be contacted by telephone, 6 months after last dose of study drug for a long-term follow-up safety survey.

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of Crohn's disease (CD) established at least 3 months prior to Screening by clinical and endoscopic evidence corroborated by a histopathology report. Cases of CD established at least 6 months prior to randomization for which a histopathology report is not available will be considered based on the weight of evidence supporting the diagnosis and excluding other potential diagnosis, and must be discussed with the sponsor on a case-by-case basis prior to randomization.
2. Has moderately to severely active CD as determined by a Crohn's Disease Activity Index (CDAI) score of 220 to 400 within 7 days prior to the first dose of study drug and 1 of the following:

   * C-reactive protein (CRP) level >2.87 mg/L during the Screening Phase, OR
   * Ileocolonoscopy with photographic documentation of a minimum of 3 nonanastomotic ulcerations (each >0.5 cm in diameter) or 10 aphtous ulcerations (involving a minimum of 10 contiguous cm of intestine) consistent with CD, within 4 months prior to randomization, OR
   * Fecal calprotectin >250 μg/g stool during the Screening Phase in conjunction with computed tomography enterography (CTE), magnetic resonance enterography (MRE), contrast enhanced small bowel radiography, or wireless capsule endoscopy revealing CD ulcerations (aphthae not sufficient), within 4 months prior to Screening
3. Has CD involvement of the ileum and/or colon, at a minimum.
4. Has extensive colitis or pancolitis of >8 years duration or limited colitis of >12 years duration must have documented evidence that a surveillance colonoscopy was performed within 12 months prior to initial screening (may be performed during Screening if not performed in previous 12 months).
5. Has a family history of colorectal cancer, personal history of increased colorectal cancer risk, age >50 years, or other known risk factor must be up-to-date on colorectal cancer surveillance (may be performed during Screening).
6. Has demonstrated an inadequate response to, loss of response to, or intolerance of at least 1 of the following agents as defined below:

   * Corticosteroids.
   * Immunomodulators.
   * Tumor necrosis factor-alpha (TNF-α) antagonists.

Exclusion Criteria:

1. Has evidence of abdominal abscess at the initial Screening Visit.
2. Has had extensive colonic resection, subtotal or total colectomy.
3. Has a history of >3 small bowel resections or diagnosis of short bowel syndrome.
4. Has had ileostomy, colostomy, known fixed symptomatic stenosis of the intestine, or evidence of fixed stenosis, or small bowel stenosis with prestenotic dilation.
5. Has had previous exposure to approved or investigational anti-integrins (e.g., natalizumab, efalizumab, etrolizumab, or AMG-181), or MAdCAM-1 antagonists, or rituximab.
6. Has used topical (rectal) treatment with 5-ASA, corticosteroid enemas/suppositories or traditional Chinese medications for CD treatment within 2 weeks of the administration of the first dose of study drug.
7. Requires currently or is anticipated to require surgical intervention for CD during the study.
8. Has a history or evidence of adenomatous colonic polyps that have not been removed.
9. Has a history or evidence of colonic mucosal dysplasia including low or high-grade dysplasia, as well as indeterminate for dysplasia.
10. Has a suspected or confirmed diagnosis of ulcerative colitis, indeterminate colitis, ischemic colitis, and radiation colitis.
11. Has evidence of treatment for C.difficile infection or other intestinal pathogen with 28 days prior to first dose of study drug.
12. Has chronic hepatitis B virus (HBV) infection or chronic hepatitis C virus (HCV) infection.
13. Has active or latent tuberculosis.
14. Has any identified congenital or acquired immunodeficiency (e.g., common variable immunodeficiency, human immunodeficiency virus [HIV] infection, organ transplantation).
15. Has any history of malignancy, except for the following: (a) adequately-treated nonmetastatic basal cell skin cancer; (b) squamous cell skin cancer that has been adequately treated and that has not recurred for at least 1 year prior to randomization; and (c) history of cervical carcinoma in situ that has been adequately treated and that has not recurred for at least 3 years prior to randomization. Participants with remote history of malignancy (e.g., >10 years since completion of curative therapy without recurrence) will be considered based on the nature of the malignancy and the therapy received and must be discussed with the sponsor on a case-by-case basis prior to randomization.
16. Has a history of any major neurological disorders, including stroke, multiple sclerosis, brain tumor, or neurodegenerative disease.
17. Has a positive progressive multifocal leukoencephalopathy (PML) subjective symptom checklist at Screening or prior to the administration of the first dose of study drug at Week 0.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2020-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director Clinical Science, Study Director — Takeda
Locations (17):
- China (17):
  - Gastroenterology, Hefei, Anhui
  - Gastroenterology, Beijing, Beijing Municipality
  - Gastroenterology, Chongqing, Chongqing Municipality
  - Gastroenterology, Fuzhou, Fujian
  - Gastroenterology, Xiamen, Fujian
  - Gastroenterology, Guangzhou, Guangdong
  - Gastroenterology, Wuhan, Hubei
  - Gastroenterology, Changsha, Hunan
  - Gastroenterology, Nanjing, Jiangsu
  - Gastroenterology, Wuxi, Jiangsu
  - Gastroenterology, Nanchang, Jiangxi
  - Gastroenterology, Changchun, Jilin
  - Gastroenterology, Shenyang, Liaoning
  - Gastroenterology, Shanghai, Shanghai Municipality
  - Gastroenterology, Chengdu, Sichuan
  - Gastroenterology, Kunming, Yunnan
  - Gastroenterology, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click on this link. — https://clinicaltrials.takeda.com/study-detail/5f6b603b4db2bf003ab4a32b?idFilter=%5B%22Vedolizumab-3034%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 27 investigative sites in China from 3 August 2017 to 14 August 2020.
Pre-assignment Details: Participants with moderately to severely active Crohn's disease were enrolled and randomized in 2:1 ratio to receive vedolizumab 300 mg or placebo in the Induction Phase of the study. Participants who achieved clinical response at Week 10 entered Maintenance Phase and continued the same study drug, placebo for every 4 weeks and vedolizumab 300 mg for every 8 weeks up to Week 58. Participants who did not achieve response received vedolizumab 300 mg every 4 weeks up to Week 58.
Period: Induction Phase (Week 0 to Week 10)
Arm/Group | Induction Phase: Placebo | Induction Phase: Vedolizumab 300 mg | Maintenance Phase: Induction Placebo to Placebo Q4W | Maintenance Phase: Induction Placebo to Vedolizumab 300 mg Q4W | Maintenance Phase: Induction Vedolizumab 300 mg to Vedolizumab 300 mg Q8W | Maintenance Phase: Induction Vedolizumab 300 mg to Vedolizumab 300 mg Q4W
Started | 71 | 144 | 0 | 0 | 0 | 0
Treated (Full Analysis Set (FAS) for the induction phase study included all randomized participants who received any amount of blinded study drug during the Induction Phase.) | 70 | 144 | 0 | 0 | 0 | 0
Completed (Completed = Participants who completed the treatment.) | 61 | 138 | 0 | 0 | 0 | 0
Not Completed | 10 | 6 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 4 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Enrolled but not Treated | 1 | 1 | 0 | 0 | 0 | 0
Period: Maintenance Phase (Week 10 to Week 60)
Arm/Group | Induction Phase: Placebo | Induction Phase: Vedolizumab 300 mg | Maintenance Phase: Induction Placebo to Placebo Q4W | Maintenance Phase: Induction Placebo to Vedolizumab 300 mg Q4W | Maintenance Phase: Induction Vedolizumab 300 mg to Vedolizumab 300 mg Q8W | Maintenance Phase: Induction Vedolizumab 300 mg to Vedolizumab 300 mg Q4W
Started | 0 | 0 | 18 | 38 | 46 | 88
Completed | 0 | 0 | 17 | 27 | 36 | 67
Not Completed | 0 | 0 | 1 | 11 | 10 | 21
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 4 | 3 | 7
Not completed — Lack of Efficacy | 0 | 0 | 1 | 3 | 3 | 4
Not completed — Reason not Specified | 0 | 0 | 0 | 4 | 4 | 10

BASELINE CHARACTERISTICS:
Population: FAS for the induction phase study included all randomized participants who received any amount of blinded study drug during the Induction Phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | Induction Phase: Placebo | Induction Phase: Vedolizumab 300 mg | Total
Number analyzed (Participants) | 70 | 144 | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.1 (8.12) | 31.1 (10.10) | 31.1 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 48 | 64
  Male | 54 | 96 | 150
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 70 | 144 | 214
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 70 | 144 | 214
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 54.61 (10.662) | 54.33 (10.388) | 54.42 (10.454)
Height [Mean (Standard Deviation); unit: cm] | 168.18 (7.785) | 166.96 (8.064) | 167.36 (7.976)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI = weight (kg)/[height (m)^2]
  kg/m^2 | 19.21 (2.978) | 19.38 (2.742) | 19.33 (2.815)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Enhanced Clinical Response in the Induction Phase at Week 10
Description: Enhanced clinical response was defined as ≥100-point decrease from Baseline in the Crohn's Disease Activity Index (CDAI) score at Week 10. A CDAI is a multi-item instrument which measures severity of active Crohn's Disease monitored over 7 days includes participant reported symptoms, physician-assessed signs, and laboratory markers. CDAI score is equal to sum of weighted scores for subjective items (number of liquid/soft stools, degree of abdominal pain, general well-being); and objective items (use of anti-diarrhoeal medication, abdominal mass, haematocrit, presence of extraintestinal manifestation, body weight). CDAI scores range approximately from 0 to 600, higher scores indicating greater disease activity.
Time Frame: Week 10
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Phase: Placebo | Induction Phase: Vedolizumab 300 mg
Number analyzed (Participants) | 70 | 144
percentage of participants | 24.3 [14.8 to 36.0] | 19.4 [13.3 to 26.9]
Statistical Analysis 1: Comparison: Induction Phase: Placebo vs Induction Phase: Vedolizumab 300 mg; Test type: Superiority; p = 0.347, Cui-Hung-Wang (CHW) test — P-value was based on CHW test, based on weighted CMH chi-square test, with stratification according to: (1)previous failure of TNF-α antagonist therapy/concomitant use of immunomodulators(Yes/No);(2)concomitant use of oral corticosteroids(Yes/No); Risk Difference (RD) = -5.2, 95% CI 2-sided [-17.2 to 6.8] — Mantel-Haenszel estimate of the treatment difference and its variance was used to calculate the 95% confidence interval for the treatment difference. Adjustment to the stratification factors was implemented

2. Secondary Outcome: Percentage of Participants With Clinical Remission in the Induction Phase at Week 10
Description: Clinical remission was defined as CDAI score of ≤150 points at Week 10. A CDAI is a multi-item instrument which measures severity of active Crohn's Disease monitored over 7 days includes participant reported symptoms, physician-assessed signs, and laboratory markers. CDAI score is equal to sum of weighted scores for subjective items (number of liquid/soft stools, degree of abdominal pain, general well-being); and objective items (use of anti-diarrhoeal medication, abdominal mass, haematocrit, presence of extraintestinal manifestation, body weight). CDAI scores range approximately from 0 to 600, higher scores indicating greater disease activity
Time Frame: Week 10
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Phase: Placebo | Induction Phase: Vedolizumab 300 mg
Number analyzed (Participants) | 70 | 144
percentage of participants | 11.4 [5.1 to 21.3] | 9.0 [4.9 to 14.9]
Statistical Analysis 1: Comparison: Induction Phase: Placebo vs Induction Phase: Vedolizumab 300 mg; Test type: Superiority; p = 0.531, Cochran-Mantel-Haenszel — P-value based on Cochran-Mantel-Haenszel, weighted CMH chi-square test, with stratification according to:(1)previous failure of TNF-α antagonist therapy/concomitant use of immunomodulators(Yes/No);(2)concomitant use of oral corticosteroids(Yes/No); Risk Difference (RD) = -2.7, 95% CI 2-sided [-11.5 to 6.0] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From first dose of the study drug up to 18 weeks after the last dose (Induction Phase: Up to Week 28; Maintenance Phase: Up to Week 78)
Description: At each visit the investigator had to document any occurrence of adverse events and clinically significant abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety Analysis Set for Induction Phase and Maintenance Phase included participants who received at least 1 dose of study drug in Induction and Maintenance Phase, respectively.
Arm/Group | Induction Phase: Placebo | Induction Phase: Vedolizumab 300 mg | Maintenance Phase: Induction Placebo to Placebo Q4W | Maintenance Phase: Induction Placebo to Vedolizumab 300 mg Q4W | Maintenance Phase: Induction Vedolizumab 300 mg to Vedolizumab 300 mg Q8W | Maintenance Phase: Induction Vedolizumab 300 mg to Vedolizumab 300 mg Q4W
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/144 | 0/18 | 0/38 | 0/46 | 1/88
Serious Adverse Events (participants affected / at risk) | 5/70 | 12/144 | 3/18 | 10/38 | 14/46 | 25/88
Other Adverse Events (participants affected / at risk) | 26/70 | 60/144 | 12/18 | 23/38 | 27/46 | 63/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Phase: Placebo (N=70) | Induction Phase: Vedolizumab 300 mg (N=144) | Maintenance Phase: Induction Placebo to Placebo Q4W (N=18) | Maintenance Phase: Induction Placebo to Vedolizumab 300 mg Q4W (N=38) | Maintenance Phase: Induction Vedolizumab 300 mg to Vedolizumab 300 mg Q8W (N=46) | Maintenance Phase: Induction Vedolizumab 300 mg to Vedolizumab 300 mg Q4W (N=88)
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 4 | 1 | 5 | 9 | 7
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1
Gastrointestinal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1
Intestinal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 1
Hyperpyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bartholin's abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3
Volvulus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ileal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Granuloma (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Anal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Mumps (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Foreign body in throat (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anal abscess (Infections and infestations) | 1 | 1 | 1 | 0 | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Phase: Placebo (N=70) | Induction Phase: Vedolizumab 300 mg (N=144) | Maintenance Phase: Induction Placebo to Placebo Q4W (N=18) | Maintenance Phase: Induction Placebo to Vedolizumab 300 mg Q4W (N=38) | Maintenance Phase: Induction Vedolizumab 300 mg to Vedolizumab 300 mg Q8W (N=46) | Maintenance Phase: Induction Vedolizumab 300 mg to Vedolizumab 300 mg Q4W (N=88)
Anaemia (Blood and lymphatic system disorders) | 6 | 8 | 2 | 2 | 6 | 10
Mouth ulceration (Gastrointestinal disorders) | 3 | 10 | 1 | 1 | 2 | 10
Pyrexia (General disorders) | 2 | 13 | 3 | 2 | 6 | 11
Protein urine present (Investigations) | 5 | 13 | 1 | 3 | 4 | 10
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 5
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 9
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 6
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 5
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 0 | 2
Nasopharyngitis (Infections and infestations) | 6 | 14 | 1 | 2 | 2 | 10
Upper respiratory tract infection (Infections and infestations) | 3 | 11 | 0 | 4 | 5 | 12
Weight decreased (Investigations) | 0 | 0 | 1 | 1 | 3 | 4
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 2 | 2 | 3
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 3 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 2 | 5
Blood urine present (Investigations) | 0 | 0 | 0 | 5 | 1 | 8
Lymphocyte count decreased (Investigations) | 7 | 8 | 2 | 3 | 4 | 3
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 2 | 1 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 3 | 3
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 2 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT03234907/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT03234907/SAP_001.pdf